CLINICAL TRIAL: NCT05881200
Title: Magnetic Mitohormesis: Effect of Magnetic Signals on Metabolic Adaptions in Type 2 Diabetes
Brief Title: Magnetic Mitohormesis: Effect of Magnetic Signals on Metabolic Adaptions in Type 2 Diabetes (MENSA-T2D)
Acronym: MENSA-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: QuantumTX Pte Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MENSA-T2D
Record Dates: First submitted 2023-04-20; First posted 2023-05-31 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Exercise; Insulin resistance; Magnetic mitohormesis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic mitohormesis (Experimental): Treatment using the BIXEPS machine
  Interventions: Device: Magnetic mitohormesis

INTERVENTIONS:
Device: Magnetic mitohormesis — The BIXEPS machine employs gentle pulsed magnetic signals specifically tuned to activate the natural "powerhouse" (mitochondria) within muscle. Brief 10-minute MM sessions with the device recreate similar biological and metabolic effects as exercise, but without physical stress or strain. It is intended to improve the strength and function of users, promoting overall fitness and well-being. Just like exercise, these effects accumulate with time.
  Subjects will receive 12 sessions of 10 minute treatments

SUMMARY:
Magnetic Mitohormesis (MM) replicates the metabolic and regenerative effects of exercise using an equipment called the BIXEPS machine, which introduces magnetic fields to the thigh muscles in a non-invasive and painless manner. Since exercise improves the blood glucose control of patients with Type 2 Diabetes Mellitus (T2DM), we believe that MM can provide the same benefits.

This single-arm pilot study investigates the effect of MM therapy on glycemic control in individuals with T2DM.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is becoming a significant health issue in the ageing Singapore population. Exercise has been shown to improve peripheral insulin sensitivity, and exercise interventions are often prescribed alongside medication to manage diabetes. However, patient compliance with diet and exercise intervention regimes can often be challenging.

Magnetic Mitohormesis (MM) is an alternative method of muscle and mitochondria activation. MM sessions are brief 10-minute weekly sessions that recreate similar biological and metabolic adaptations as exercise but without physical stress or strain. MM can be easily applied to any age group while seated and without limitations on users' physical aptitude.

Having MM as an adjunct therapy to exercise and drug interventions could improve glycaemic control in T2DM patients, especially amongst the ageing population and those with less exercise capacity.

This single-arm pilot study investigates the effect of MM therapy on glycemic control in individuals with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years
2. T2DM of at least 6 months duration
3. HbA1c between 7.0% - 10.0% (most recent 3-months prior to enrolment)
4. Body Mass Index (BMI) between 23.0 and 32.5 kg/m2
5. Able to ambulate independently
6. Willing and able to give written informed consent

Exclusion Criteria:

1. Presence of any conditions contraindicated for PEMF exposures (e.g. active electronic implants, pregnancy, pacemakers, implantable defibrillators)
2. Medical advice against physical activity
3. Chest pain when performing physical activity
4. Chest pain at rest
5. BP > 180/90 mmHg
6. Women who are lactating, pregnant or considering pregnancy
7. Cancer not in remission or receiving active cancer treatment
8. Current participation in another clinical trial
9. Systemic steroid usage (eg. prednisolone, hydrocortisone, cortisone, dexamethasone)
10. Uncontrolled thyroid disease
11. Significant alcohol intake (> 1 unit per day for women and > 2 units per day for men)
12. Any factors likely to limit adherence to study protocol (e.g. dementia; alcohol or substance abuse; history of unreliability in medication taking or appointment keeping; significant concerns about participation in the study from spouse, significant other or family members)
13. Anticipated surgery or changes in diabetes medications during the study duration
14. History of severe hypoglycaemia in the recent 3 months
15. Have used the MM device in the past 3 months
16. Had a recent surgical procedure in the last 6 months, where muscle activation can interfere with the healing response

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1C | 12 weeks
  Change in glycemic control
Change in insulin resistance | 12 weeks
  Change in Homeostatic Model Assessment for Insulin Resistance index

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chang Tan, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Png ME, Yoong J, Phan TP, Wee HL. Current and future economic burden of diabetes among working-age adults in Asia: conservative estimates for Singapore from 2010-2050. BMC Public Health. 2016 Feb 16;16:153. doi: 10.1186/s12889-016-2827-1. PMID 26880337
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement. Diabetes Care. 2010 Dec;33(12):e147-67. doi: 10.2337/dc10-9990. PMID 21115758